CLINICAL TRIAL: NCT05118386
Title: A Phase 1 Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of RSM01, a Monoclonal Antibody Targeting Respiratory Syncytial Virus, in Healthy Adults
Brief Title: Safety, Tolerability, and Pharmacokinetics of RSV Monoclonal Antibody RSM01 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gates Medical Research Institute (Other)
Collaborators: PPD Phase I Clinic - Orlando (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gates MRI-RSM01-101
Record Dates: First submitted 2021-10-06; First posted 2021-11-12 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2023-12

CONDITIONS: RSV Infection
Keywords: Monoclonal antibody
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled study of RSM01. The study was conducted in 2 parts: A Dose Escalation Phase (28 participants) with 4 dosing cohorts, followed by an Expansion Phase (28 participants) with a single cohort.
Who Masked: Participant, Investigator
Masking Description: Participants and all study personnel were blinded to the randomization. Authorized study site personnel would administer doses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RSM01 (Experimental): Participants were randomized to receive different dose levels of RSM01. Participants were randomized in a ratio of 6:1 where for every 6 participants received active drug (RSM01), 1 participant received Placebo.
  Interventions: Drug: RSM01
- Placebo (Placebo Comparator): Participants received Placebo matched to RSM01.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RSM01 — Cohort 1: RSM01 300 mg IV
  Cohort 2: RSM01 300 mg IM
  Cohort 3: RSM01 1000 mg IV
  Cohort 4: RSM01 3000 mg IV
  Cohort 5: RSM01 600 mg IM
  Arms: RSM01
Other: Placebo — Cohort 1: Placebo IV
  Cohort 2: Placebo IM
  Cohort 3: Placebo IV
  Cohort 4: Placebo IV
  Cohort 5: Placebo IM
  Arms: Placebo

SUMMARY:
Gates MRI-RSM01-101 was a Phase 1, randomized, double-blind, placebo-controlled, dose-escalation study to evaluate the safety and tolerability, pharmacokinetics, occurrence of Anti-drug antibody (ADA), and assessment of neutralizing antibody against RSV after administration of single intravenous or intramuscular doses of RSM01 to healthy adults.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is the most common cause of lower respiratory tract infection (LRTI) among infants and young children, resulting in annual epidemics worldwide.

RSM01, a monoclonal antibody targeting RSV, may potentially provide an effective method to protect infants from RSV disease based on its potency and an extended half-life that is expected to support once-per-RSV-season administration.

This study was a first-in-human evaluation of RSM01 in healthy male and female adults with the goal of characterizing the safety and tolerability of a range of single doses of RSM01 to enable determination of appropriate dose(s) to be administered to infants in a future study. Enrollment was planned at a single study center in the United States. 56 participants were enrolled; 48 participants received RSM01 and 8 participants received Placebo. Participants were followed for approximately 5 months (151 days) after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 49 years of age (inclusive), at the time of signing the informed consent.
2. Participant is healthy as determined by medical evaluation including medical history, physical examination and laboratory tests.
3. Body mass index (BMI) 18 to 29.9 kg/m2 (inclusive)
4. Both males and females are eligible to participate. Female participants must not be pregnant, breastfeeding, or attempting to become pregnant for 28 days prior to screening and throughout the duration of the study. Females must be willing to comply with protocol-specified contraception for the duration of their participation in the study and for 90 days following the completion of the study. Male participants with partners of childbearing potential must be willing to comply with protocol specific contraception for the duration of their participation in the study and for 90 days following the completion of the study. Males must also agree to refrain from sperm donation for at least 90 days after they complete the study.
5. Participant must be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol
6. Participant agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to relocate from the study area for the duration of the study.

Exclusion Criteria:

1. Acute illness and/or body temperature ≥37.5°C or ≥99.5°F on Study Day 1. NOTE: This is a temporary exclusion for which the participant may be re-evaluated
2. Evidence and/or history of clinically significant medical condition(s) as judged by the investigator, including malignancies, diabetes mellitus, and unstable or uncontrolled hypertension
3. History of any autoimmune disease or immune deficiency or other impairment to the immune system, including but not limited to HIV, autoimmune conditions, or immunosuppressive therapy. Note: history of Hashimoto's thyroiditis is not an exclusion criterion
4. History of anaphylaxis
5. Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the participant will comply with the protocol
6. Receiving or plans to receive any medications or other therapies that may impact the immune system such as allergy injections, interferon, immunomodulators, cytotoxic drugs or other drugs known to be frequently associated with major organ toxicity within 90 days prior to Day 1
7. Received any vaccination (including COVID-19 vaccine) within the 15 days before Day 1 or plans to receive a dose of any vaccine during the 15-day period following Day 1
8. Receiving or plans to receive immunosuppressive agents including systemic steroids within 90 days prior to Day 1 (individuals using inhaled or topical corticosteroids, prednisone (or equivalent) dose of ≤ 20 mg/day for ≤ 14 days, and intra-articular corticosteroids are permitted)
9. Received or donated blood or blood products within 90 days prior to Day 1 or plans to receive or donate during the study period
10. Received or plans to receive antibody or biologic therapy within 180 days prior to Day 1 or any time during the study period, whether licensed or investigational (e.g., immunoglobulin products, monoclonal antibodies, or antibody fragments)
11. Participation in an interventional clinical trial and/or receipt of any investigational drug within 30 days or 5 half-lives of the investigational drug before the first day of study drug dosing in this study, whichever is longer.
12. Concurrent enrollment in another interventional study
13. Previously participated and received study intervention in the current study
14. Female participants: positive serum pregnancy test
15. Safety laboratory values outside of normal range, for age and sex that are suggestive of a disease state (Grade 1 abnormalities will not lead to exclusion if the investigator considers them not clinically significant.)
16. Urinalysis abnormality greater than Grade 1 (with the exception of hematuria in a menstruating female), or urinalysis abnormality judged clinically significant by the investigator
17. Clinically significant ECG abnormalities
18. Reactive HIV antibody testing
19. Current hepatitis B and/or hepatitis C infection
20. Positive urine drug screen at screening or Day -1 (with the exception of prescribed drugs)
21. History of allergy or hypersensitivity to the study drug, excipients or related substances
22. Female participants with any one of the following conditions: currently pregnant or lactating/nursing; has positive serum pregnancy test during the Screening Phase, planning a pregnancy within 1 year after first dose of study drug
23. Acting as study personnel or immediate family members (brother, sister, child, parent) or the spouse/partner of study personnel

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gates MRI, Study Director — Gates Medical Research Institute
Locations (1):
- PPD Phase I Clinic - Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized or deidentified, as appropriate, participant level data may be shared with external researchers in accordance with the trial participants' written and executed informed consent document and any local or applicable regulations on data sharing. Qualified researchers may submit a request for anonymized or de-identified participant level data along with a research proposal to Gates MRI for review. A data sharing agreement must be in place before any clinical trial data are shared. There are additional circumstances that may prevent the sharing of data with external researchers, including but not limited to contractual obligations to existing partners and any restrictions imposed by regulatory bodies.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] White JT, Terstappen J, Levi M, Radivojevic A, Noble R, Anderson AB, Wise-Blackman G, Dunne MW. Replacing serum with dried blood microsampling for pharmacokinetics, viral neutralisation and immunogenicity bioanalysis supporting future paediatric development of RSM01, a candidate respiratory syncytial virus neutralising monoclonal antibody. BMC Infect Dis. 2024 Dec 18;24(1):1403. doi: 10.1186/s12879-024-10196-4. PMID 39696004
- [Derived] Bonavia A, Levi M, Rouha H, Badarau A, Terstappen J, Watson S, Anderson AB, White JT, Ananworanich J, Taylor D, Radivojevic A, Shaffer M, Stamm LM, Dunne MW. RSM01, a novel respiratory syncytial virus monoclonal antibody: preclinical characterization and results of a first-in-human, randomised clinical trial. BMC Infect Dis. 2024 Dec 3;24(1):1378. doi: 10.1186/s12879-024-10120-w. PMID 39627701
- [Derived] Terstappen J, Delemarre EM, Versnel A, White JT, Derrien-Colemyn A, Ruckwardt TJ, Bont LJ, Mazur NI. RSV Neutralizing Antibodies in Dried Blood. J Infect Dis. 2024 Jul 25;230(1):e93-e101. doi: 10.1093/infdis/jiad543. PMID 39052716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in United States
Pre-assignment Details: The study was conducted in 2 parts: Dose Escalation Phase followed by an Expansion Phase. Participants were randomized 6:1 to RSM01 or Placebo in each dose cohort. Results are presented by intervention.
Groups:
- RSM01 300 Milligrams (mg) Intravenous (IV): Within the RSM01 300 mg IV dose cohort, participants were randomized to receive RSM01 300 mg IV
- RSM01 300 mg Intramuscular (IM): Within the RSM01 300 mg IM dose cohort, participants were randomized to receive RSM01 300 mg IM
- RSM01 1000 mg IV: Within the RSM01 1000 mg IV dose cohort, participants were randomized to receive RSM01 1000 mg IV
- RSM01 3000 mg IV: Within the RSM01 3000 mg IV dose cohort, participants were randomized to receive RSM01 3000 mg IV
- RSM01 600 mg IM: Within the RSM01 600 mg IM dose cohort, participants were randomized to receive RSM01 600 mg IM
- Placebo: Participants randomized to Placebo within the dose cohorts are pooled.
Period: Dose Escalation Phase (Day 1 to Day 151)
Arm/Group | RSM01 300 Milligrams (mg) Intravenous (IV) | RSM01 300 mg Intramuscular (IM) | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM | Placebo
Started | 6 | 6 | 6 | 6 | 0 | 4
Completed | 6 | 6 | 6 | 4 | 0 | 4
Not Completed | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 0
Period: Dose Expansion Phase (Day 1 to Day 151)
Arm/Group | RSM01 300 Milligrams (mg) Intravenous (IV) | RSM01 300 mg Intramuscular (IM) | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM | Placebo
Started | 0 | 0 | 0 | 0 | 24 | 4
Completed | 0 | 0 | 0 | 0 | 23 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Unspecified Reason Not Completed | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: included all participants who received the study treatment.
Groups:
- RSM01 300 mg IV: Within the RSM01 300 mg IV dose cohort, participants were randomized to receive RSM01 300 mg IV
- RSM01 300 mg IM: Within the RSM01 300 mg IM dose cohort, participants were randomized to receive RSM01 300 mg IM
- Total: Total of all reporting groups
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24 | 8 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.2 (4.26) | 30.7 (9.40) | 31.5 (8.76) | 27.5 (9.54) | 34.1 (8.69) | 30.9 (5.33) | 31.6 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 5 | 2 | 11 | 5 | 27
  Male | 5 | 3 | 1 | 4 | 13 | 3 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 4 | 6 | 12 | 2 | 29
  Not Hispanic or Latino | 4 | 3 | 2 | 0 | 12 | 6 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 2 | 2 | 0 | 6 | 3 | 14
  White | 4 | 4 | 3 | 5 | 16 | 5 | 37
  More than one race | 1 | 0 | 1 | 0 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unsolicited Treatment Emergent Adverse Events (TEAEs) Through Day 151
Description: A TEAE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A memory aid was utilized by participants to collect unsolicited TEAEs beginning at discharge from the clinic, through Day 151. Participants were instructed to record unsolicited TEAEs whenever they occurred, recording such TEAEs on the memory aid. The memory aids were collected and reviewed by site staff at each subsequent visit through the end of the study. Number of participants with unsolicited TEAEs through Day 151 has been presented.
Time Frame: Day 1 through Day 151
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24 | 8
Participants | 1 | 2 | 3 | 3 | 3 | 2

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and AE of Special Interest (AESIs) Through Day 151
Description: An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. AESIs were defined as events of potential immunologic etiology, including immune-related AEs (irAEs). Number of participants with SAEs and AESIs through Day 151 has been presented.
Time Frame: Day 1 through Day 151
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24 | 8
Participants
  SAEs | 0 | 0 | 0 | 0 | 0 | 0
  AESI | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Solicited Systemic AEs for 7 Days After Dose Administration
Description: Solicited systemic AEs were defined events that participants were specifically asked about and which were noted by participants in the diary card. Systemic solicited AEs included fever, headache, tiredness, joint pain, muscle pain, nausea, vomiting and diarrhea. Number of participants with solicited systemic AEs for 7 days after dose administration has been presented.
Time Frame: Through Day 7
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- RSM01 3000 mg IV: Within the RSM01 1000 mg IV dose cohort, participants were randomized to receive RSM01 3000 mg IV
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24 | 8
Participants
  Fever | 0 | 0 | 0 | 0 | 0 | 1
  Headache | 0 | 2 | 2 | 0 | 1 | 0
  Tiredness | 0 | 0 | 0 | 0 | 2 | 0
  Joint pain | 0 | 0 | 0 | 0 | 0 | 0
  Muscle pain | 0 | 0 | 0 | 0 | 0 | 0
  Nausea | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Solicited Local AEs for Injection Site Reactions for 7 Days After Intramuscular Dose Administration
Description: Solicited local AEs were defined events that participants were specifically asked about and which were noted by participants in the diary card. Solicited local AEs for injection site reactions included AEs include pain, redness and swelling. Number of participants with solicited local AEs for injection site reactions for 7 days after intramuscular dose administration has been presented
Time Frame: Up to Day 7
Population: Safety Population. Data has been presented only for participants who received RSM01 and placebo intramuscularly.
Measure: Count of Participants; unit: Participants
Arm/Group | RSM01 300 mg IM | RSM01 600 mg IM | Placebo
Number analyzed (Participants) | 6 | 24 | 5
Participants
  Pain | 0 | 2 | 0
  Redness | 0 | 2 | 0
  Swelling | 0 | 1 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Hematology Assessments of Grade 1 and Above Through Day 151
Description: Blood samples were collected for the assessment of hemoglobin, platelets, leukocytes, neutrophils and lymphocytes. Laboratory grades were evaluated using the Food and Drug administration (FDA) Toxicity Grading Scale with grading as: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening or disabling. Number of participants with clinically significant hematology assessments of Grade 1 and above has been presented.
Time Frame: Through Day 151
Population: Safety Population. Only those participants with data available at specified time points has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 23 | 8
Participants
  Hemoglobin: Grade 1 | 0 | 0 | 1 | 0 | 0 | 0
  Hemoglobin: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils: Grade 1 | 0 | 0 | 0 | 0 | 2 | 2
  Neutrophils: Grade 2 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophils: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Clinical Chemistry Assessments of Grade 1 and Above Through Day 151
Description: Blood samples were collected for the assessment of Alanine Aminotransferase, Aspartate Aminotransferase, Alkaline Phosphatase, Bilirubin, Gamma Glutamyl Transferase, Creatinine, Urea nitrogen, Glucose, Albumin, Sodium and Potassium. Laboratory grades were evaluated using the FDA Toxicity Grading Scale with grading as: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening or disabling. Number of participants with clinically significant clinical chemistry assessments of Grade 1 and above has been presented.
Time Frame: Through Day 151
Population: Safety Population. Only those participants with data available at specified time points has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 23 | 8
Participants
  Alanine Aminotransferase: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Grade 1 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Urea nitrogen: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urea nitrogen: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Urea nitrogen: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Urea nitrogen: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose: Grade 1 | 1 | 0 | 0 | 0 | 0 | 0
  Glucose: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Area Under the Capillary Blood-concentration Time Curve From Zero to Infinity (AUC 0-infinity) After Administration of RSM01
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of RSM01. PK parameters were analyzed using standard non-compartmental analysis. AUC(0-infinity) in participants with AUC extrapolation exceeding 20% was deemed unreliable in the terminal phase and thus omitted from the summary statistics.
Time Frame: Day 151
Population: Pharmacokinetic (PK) population: included all participants who received the study intervention. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter (h*ng/mL)
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM
Number analyzed (Participants) | 1 | 2 | 2 | 1 | 1
Hours*nanograms per milliliter (h*ng/mL) | 25700000 (NA) — Not applicable (NA) indicates geometric coefficient of variation could not be calculated as a single participant was analyzed. | 25300000 (23.6) | 239000000 (26.4) | 1010000000 (NA) — Not applicable (NA) indicates geometric coefficient of variation could not be calculated as a single participant was analyzed. | 106000000 (NA) — Not applicable (NA) indicates geometric coefficient of variation could not be calculated as a single participant was analyzed.

8. Secondary Outcome: Day 91 Capillary Blood-concentration (CD91) After Administration of RSM01
Description: Blood samples were collected at indicated time points for PK analysis of RSM01. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Day 91
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Nanograms per milliliter (ng/mL) | 14500 (83.5) | 8020 (209.6) | 63400 (38.8) | 196000 (25.9) | 27600 (76.7)

9. Secondary Outcome: Day 91 Area Under the Capillary Blood-concentration Time Curve (AUC 0-D91) After Administration of RSM01
Description: as for outcome 8
Time Frame: Day 91
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter (h*ng/mL)
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Hours*nanograms per milliliter (h*ng/mL) | 50900000 (42.0) | 40600000 (44.3) | 207000000 (22.8) | 549000000 (17.3) | 85400000 (39.3)

10. Secondary Outcome: Day 151 Capillary Blood-concentration (CD151) After Administration of RSM01
Description: as for outcome 8
Time Frame: Day 151
Population: PK population. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 23
Nanograms per milliliter (ng/mL) | 13500 (13.4) | 12100 (8.2) | 36800 (58.8) | 105000 (32.7) | 17900 (76.8)

11. Secondary Outcome: Day 151 Area Under the Capillary Blood-concentration Time Curve (AUC 0-D151) After Administration of RSM01
Description: as for outcome 8
Time Frame: Day 151
Population: PK population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter (h*ng/mL)
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM
Number analyzed (Participants) | 6 | 5 | 6 | 4 | 23
Hours*nanograms per milliliter (h*ng/mL) | 68700000 (53.8) | 48400000 (69.3) | 278000000 (27.5) | 813000000 (22.9) | 114000000 (48.3)

12. Secondary Outcome: Maximum Capillary Blood Concentration (Cmax) After Administration of RSM01
Description: as for outcome 8
Time Frame: Day 151
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Nanograms per milliliter (ng/mL) | 62200 (20.3) | 31500 (17.6) | 264000 (18.2) | 652000 (13.8) | 56400 (23.9)

13. Secondary Outcome: Minimum Capillary Blood Concentration (Cmin) After Administration of RSM01
Description: as for outcome 8
Time Frame: Day 151
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (Ng/mL)
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Nanograms per milliliter (Ng/mL) | 13500 (13.4) | 3670 (68.9) | 36100 (56.7) | 127000 (38.7) | 18700 (78.5)

14. Secondary Outcome: Time to Maximum Capillary Blood-concentration (Tmax) After Administration of RSM01
Description: as for outcome 8
Time Frame: Day 151
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Hours | 1.300 [1.25 to 9.28] | 140.458 [121.35 to 168.88] | 1.808 [1.75 to 1.97] | 2.208 [2.18 to 10.17] | 193.508 [165.77 to 695.38]

15. Secondary Outcome: Apparent Terminal Half-Life After Administration of RSM01
Description: Blood samples were collected at indicated time points for PK analysis of RSM01. PK parameters were analyzed using standard non-compartmental analysis. Apparent terminal half-life in participants with AUC extrapolation exceeding 20% was deemed unreliable in the terminal phase and thus omitted from the summary statistics.
Time Frame: Day 151
Population: PK population. Only those participants with data available at the specified data points were analyzed
Measure: Median (Full Range); unit: Hours
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM
Number analyzed (Participants) | 1 | 2 | 2 | 1 | 1
Hours | 653 [653 to 653] | 439 [438 to 440] | 1310 [1220 to 1400] | 1060 [1060 to 1060] | 1480 [1480 to 1480]

16. Secondary Outcome: Total Body Clearance (CL) After Intravenous Dose Administration of RSM01
Description: Blood samples were collected at indicated time points for PK analysis of RSM01. PK parameters were analyzed using standard non-compartmental analysis. CL post intravenous administration in participants with AUC extrapolation exceeding 20% was deemed unreliable in the terminal phase and thus omitted from the summary statistics.
Time Frame: Day 151
Population: PK population. Only those participants with data available at the specified data points were analyzed. Data has been presented only for participants who received RSM01 intravenously
Measure: Mean (Standard Deviation); unit: Milliliter per hour (mL/h)
Arm/Group | RSM01 300 mg IV | RSM01 1000 mg IV | RSM01 3000 mg IV
Number analyzed (Participants) | 1 | 2 | 1
Milliliter per hour (mL/h) | 11.7 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 4.25 (1.09) | 2.98 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.

17. Secondary Outcome: Apparent Total Body Clearance (CL) After Intramuscular Dose Administration of RSM01
Description: Blood samples were collected at indicated time points for PK analysis of RSM01. PK parameters were analyzed using standard non-compartmental analysis. Total body CL post intramuscular administration in participants with AUC extrapolation exceeding 20% was deemed unreliable in the terminal phase and thus omitted from the summary statistics.
Time Frame: Day 151
Population: PK population. Only those participants with data available at the specified data points were analyzed. Data has been presented only for participants who received RSM01 intramuscularly.
Measure: Mean (Standard Deviation); unit: Milliliter per hour (mL/h)
Arm/Group | RSM01 300 mg IM | RSM01 600 mg IM
Number analyzed (Participants) | 2 | 1
Milliliter per hour (mL/h) | 12.0 (2.77) | 5.68 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed

18. Secondary Outcome: Volume of Distribution (Vz) After Intravenous Dose Administration of RSM01
Description: Blood samples were collected at indicated time points for PK analysis of RSM01. PK parameters were analyzed using standard non-compartmental analysis. Vz post intravenous administration in participants with AUC extrapolation exceeding 20% was deemed unreliable in the terminal phase and thus omitted from the summary statistics.
Time Frame: Day 151
Population: as for outcome 16
Measure: Median (Standard Deviation); unit: Milliliter (mL)
Arm/Group | RSM01 300 mg IV | RSM01 1000 mg IV | RSM01 3000 mg IV
Number analyzed (Participants) | 1 | 2 | 1
Milliliter (mL) | 11000 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 7920 (1310) | 4550 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.

19. Secondary Outcome: Apparent Volume of Distribution (Vz) After Intramuscular Dose Administration of RSM01
Description: Blood samples were collected at indicated time points for PK analysis of RSM01. PK parameters were analyzed using standard non-compartmental analysis. Vz post intramuscular administration in participants with AUC extrapolation exceeding 20% was deemed unreliable in the terminal phase and thus omitted from the summary statistics.
Time Frame: Day 151
Population: as for outcome 17
Measure: Median (Standard Deviation); unit: Milliliter (mL)
Arm/Group | RSM01 300 mg IM | RSM01 600 mg IM
Number analyzed (Participants) | 2 | 1
Milliliter (mL) | 7610 (1740) | 12200 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed

20. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADAs) at Baseline and Post-Baseline Through Day 151 Following RSM01 Administration
Description: Whole blood samples in serum separator tubes and volumetric absorptive microsampling (VAMS) samples were collected for detection of ADAs against RSM01 in serum and capillary blood, respectively. The detection of ADA to RSM01 was performed using a validated immunoassay method with tiered testing of screening, confirmatory, and titration. Number of participants with positive ADAs at Baseline and post-Baseline through Day 151 following RSM01 administration has been presented.
Time Frame: Baseline (Day 1) and post-Baseline through Day 151
Population: Immunogenicity Population: all participants who received the study intervention and have at least one valid ADA result
Measure: Count of Participants; unit: Participants
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24 | 8
Participants
  Baseline | 0 | 0 | 1 | 0 | 0 | 0
  Post-Baseline Through Day 151 | 0 | 0 | 2 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through Day 151
Description: Safety population defined as all participants who received the study treatment.
Arm/Group | RSM01 300 mg IV | RSM01 300 mg IM | RSM01 1000 mg IV | RSM01 3000 mg IV | RSM01 600 mg IM | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/24 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/24 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 3/6 | 3/6 | 3/24 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSM01 300 mg IV (N=6) | RSM01 300 mg IM (N=6) | RSM01 1000 mg IV (N=6) | RSM01 3000 mg IV (N=6) | RSM01 600 mg IM (N=24) | Placebo (N=8)
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Bartholinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT05118386/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT05118386/SAP_001.pdf